CLINICAL TRIAL: NCT02463838
Title: San Francisco Health Plan Care Support Intervention: A Randomized Trial
Brief Title: San Francisco Health Plan Care Support Trial
Acronym: SFHP_CBCM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco Health Plan (Unknown); California Health Facilities Financing Authority (CHFFA) (Other Government)
Responsible Party: Principal Investigator, Maria Raven, MD, Assistant Professor of Emergency Medicine, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 14-14737
Record Dates: First submitted 2015-05-27; First posted 2015-06-04 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Case Management; Managed Care Program
Keywords: Medi-Cal; Health Plan; Frequent Users; Heavy users; Care Coordination; Managed Care; Case Management; Mental Health; Substance Use; Emergency Department
MeSH Terms: conditions — Psychological Well-Being; Substance-Related Disorders; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Care Support Intervention (Experimental): Eligible members are assigned a CareSupport Coordinator who carries a caseload of 25-35 members. A team of 5 Coordinators is supervised by a master's level Social Worker. Community Coordinators work with members to conduct standardized assessments to develop a Care Plan shared with other providers within and outside of SFHP. Coordinators provide members advocacy and navigation across systems of care, to improve coordination focus on treatment goals. Coordinator focus on prevention and early intervention around disease management, advocacy, appointment reminders and accompaniment, home visits, and regular communication with primary care and other providers. Coordinators are encouraged to be accountable for coordinating and following through on all aspects of a member's needs.
  Interventions: Other: Care Support Intervention
- Usual Care (No Intervention): All eligible SFHP members randomized to usual care will receive medical and health plan by virtue of enrollment in the SFHP and Medi-Cal. Services include assignment to a primary care physician and access to all services available through Medi-Cal in the county of San Francisco.

INTERVENTIONS:
Other: Care Support Intervention — Case management and care coordination intervention delivered in person to SFHP members who are frequent users of emergency department and inpatient hospital services.
  Arms: Care Support Intervention

SUMMARY:
This study will expand and evaluate an existing pilot program to improve care for frequent users of acute emergency and inpatient services by providing care coordination and management for eligible San Francisco Health Plan members. SF Health Plan's Community-Based Care Management pilot program ("Program") known as "CareSupport" serves vulnerable SF Health Plan members who are high utilizers of hospital inpatient and emergency departments and at extremely high risk for mortality and morbidity due to factors such as housing instability, mental illness, and addiction. Care managers, called community coordinators, are trained bachelor-level social workers or outreach workers and each have a panel of 30-35 members who they directly engage in the community where the members tend to live or congregate (shelters, bus stops, coffee shops, community agencies, and by cell phone) to help them improve their health and navigate through the health care and social services systems. The number of San Francisco Health Plan members who would be eligible for Care Support services far outstrips the capacity the San Francisco Health Plan to provide these additional services, and the investigators will thus evaluate the intervention using a randomized trial design.

DETAILED DESCRIPTION:
Purpose: The purpose of the CareSupport intervention is to coordinate often-fragmented care for SFHP members with heavy use of acute health care services, reducing cost of care for the San Francisco safety net (the San Francisco Department of Health and San Francisco General Hospital) while increasing use of sustaining services including primary care.

The Program: The San Francisco Health Plan (SFHP) CareSupport program identifies high-utilizing SFHP members with high risk for mortality and morbidity due to factors that complicate underlying illness and care seeking patterns. These factors include housing instability, behavioral health issues, and complex medical illness. This population's medical, behavioral and social needs are not met by the existing delivery system, and while many issues they face may not be traditionally perceived as health care, they do impact this vulnerable population's health and care seeking patterns greatly.

CareSupport Community Coordinators each carry a caseload of 25-35 eligible members identified based on health services use in the prior 12 months. Each team of 5 Coordinators is supervised by a skilled master's level Social Worker. Community Coordinators outreach to eligible patients and conduct detailed assessments in order to develop a Care Plan that is then shared with other providers within and outside of SFHP. Community Coordinators provide patient-centered, community-based advocacy and navigation across systems of care, to improve coordination and unify health and treatment goals. The CareSupport program incorporates a focus on prevention and early intervention within a continuum of quality health care that includes disease management, advocacy, appointment reminders and accompaniment, home visits, and regular communication with primary care and other providers. Community Coordinators are accountable for coordinating and following through on all aspects of a member's needs, and their duties are as variable as reminder calls, accompaniment to medical appointments, assistance with housing placement, and help obtaining food and other services. Twice weekly team meetings involve complex case reviews and program troubleshooting as well as mini trainings led by social work supervisors. The staff is trained in trauma-informed care, motivational interviewing, harm reduction, and other areas of relevance to the intervention target population.

The investigators' composed of 3 groups of SFHP members, all of whom are heavy users of health care services: 1) members with a minimum of 2 hospitalizations in the year before enrollment 2) members with 5 ED visits and 1 hospitalization in the year before enrollment, and 3) members with 6 or more ED visits in the year before enrollment in the investigators' program.

The current CareSupport staff does not have the capacity to serve all SFHP members who are eligible for CareSupport. The investigators propose to ethically allocate limited resources and evaluate the impact of CareSupport using a randomly selected comparison group of non-enrolled, CareSupport eligible SFHP members.

Randomization

Randomization process: First, eligible members will be rank ordered by descending age, then based first on number of hospital admissions in the prior year, and finally by number of ED visits in the prior year. SFHP members falling into the CareSupport target population based on their utilization in the prior 12 months will be assigned using a standard "every other" technique to either the CareSupport program (the intervention) or to the comparison group that will not be offered enrollment. This technique will result in a "member pair," where one member from the pair will be randomly assigned to the CareSupport intervention and one member of the pair will be randomly assigned to the comparison group. For the purposes of the evaluation, the member pair will share the same engagement date (see below).

The investigators will use an intention to treat framework: all SFHP members assigned to CareSupport or the comparison group will remain in those groups for the analysis.

Outcomes and Evaluation Methods As mentioned above, SFHP has enrollment, demographic and encounter/claims data for all SFHP members and these data will be used to conduct the investigators' analysis. The investigators' primary outcomes can be tracked based on administrative encounter data, and will include member services use across San Francisco rather than being limited to a single hospital or small network of clinics.

A central goal of the investigators' evaluation is to determine whether the CareSupport demonstration project generates more savings to the delivery system than it costs to implement and sustain. The ability of the CareSupport program to succeed in this goal will help determine whether it is sustainable and exportable to other sites. The investigators anticipate that the CBCM model will produce cost-savings both by employing less expensive, more appropriately-trained staff, as well as by connecting vulnerable members more effectively to primary and preventive care, and social and behavioral resources, thereby reducing their use of acute care.

ELIGIBILITY:
Inclusion Criteria:

To be eligible, SFHP members must have one of three health service use patterns in the prior 12 months:

* 2 or more hospital admissions
* 5 ED visits and 1 hospital admission
* 6 or more ED visits
* Must be aged 18 or older

Exclusion Criteria:

* Under age 18
* Not a SFHP member

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
ED visits | 9-18 months
  Difference in the number of ED visits comparing intervention and usual care groups
Hospital admissions | 9-18 months
  Difference in the number of hospital admissions comparing intervention and usual care groups
Hospital bed days | 9-18 months
  Difference in the number of hospital bed days comparing intervention and usual care groups

SECONDARY OUTCOMES:
Primary care visits | 9-18 months
  Difference in the number of primary care visits comparing intervention and usual care groups
Cost of health care services | 9-18 months
  Difference in costs associated with ED visits, hospital admissions, and primary care visits comparing intervention and usual care groups, using standard Medi-Cal reimbursement rates
Net program costs | 9-18 months
  Comparative cost analysis that examines differences in Medi-Cal reimbursements in comparison to SFHP program costs (e.g. staffing, overhead). we plan to track not only the health service use costs outlined above (by assigning standard Medi-Cal reimbursement rates to each service), but also costs related to the CareSupport program such as staffing costs, supplies, and transportation via a comprehensive economic analysis.
Mental health | Baseline, 6 month follow-up, 12 month follow up if still enrolled
  Depression will be evaluated for the intervention group only, and will include depression based on the PHQ-2. Changes in scores will be assessed at baseline and 6-month follow-up as a standard part of the CareSupport assessment and follow-up process conducted by the CareSupport Community Coordinators.
Patient satisfaction | Baseline, 6 month follow-up, 12 month follow up if still enrolled
  Satisfaction will be evaluated for the intervention group only, and will include depression based on the PHQ-9. Changes in scores will be assessed at baseline and 6-month follow-up as a standard part of the CareSupport assessment and follow-up process conducted by the CareSupport Community Coordinators.
Self-reported health | Baseline, 6 month follow-up, 12 month follow up if still enrolled
  Self reported health will be evaluated for the intervention group only and will include a question from the SF-8.

CONTACTS AND LOCATIONS:
Locations (1):
- San Francisco Health Plan, San Francisco, California, United States